CLINICAL TRIAL: NCT00862459
Title: Multi-center, Double-blind, Randomized, Controlled, Parallel Group, Dose Comparison Study With Corresponding Blinded Image Evaluation Following a Single Intravenous Injection of Three Different Doses of Gadobutrol 1.0 Molar (Gadavist) in Patients With Known or Suspected Focal Blood Brain Barrier Disturbances and/or Abnormal Vascularity of the Central Nervous System
Brief Title: Dose Finding Study of Gadavist in Central Nervous System (CNS) Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 91400; 308200 (Other: company internal)
Record Dates: First submitted 2008-11-26; First posted 2009-03-17 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Brain Diseases; Spinal Cord Diseases
Keywords: Contrast Agents
MeSH Terms: conditions — Brain Diseases; Spinal Cord Diseases | interventions — gadobutrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participant received one dose of 0.03 mmol/kg BW of Gadobutrol and one dose of 0.1 mmol/kg body weight (BW) of OptiMARK. The order in which the participants received Gadobutrol and OptiMARK was randomized. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
  Interventions: Drug: Gadobutrol~0.03 mmol/kg BW (Gadavist, Gadovist, BAY86-4875); Drug: OptiMARK~0.1 mmol/kg BW
- Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participant received one dose of 0.1 mmol/kg BW of Gadobutrol and one dose of 0.1 mmol/kg BW of OptiMARK. The order in which the participants received Gadobutrol and OptiMARK was randomized. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
  Interventions: Drug: Gadobutrol~0.1 mmol/kg BW (Gadavist, Gadovist, BAY86-4875); Drug: OptiMARK~0.1 mmol/kg BW
- Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participant received one dose of 0.3 mmol/kg BW of Gadobutrol and one dose of 0.1 mmol/kg BW of OptiMARK. The order in which the participants received Gadobutrol and OptiMARK was randomized. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
  Interventions: Drug: Gadobutrol~0.3 mmol/kg BW (Gadavist, Gadovist, BAY86-4875); Drug: OptiMARK~0.1 mmol/kg BW

INTERVENTIONS:
Drug: Gadobutrol~0.03 mmol/kg BW (Gadavist, Gadovist, BAY86-4875) — Participant received one dose of 0.03 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
  Arms: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875)
Drug: Gadobutrol~0.1 mmol/kg BW (Gadavist, Gadovist, BAY86-4875) — Participant received one dose of 0.1 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
  Arms: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875)
Drug: Gadobutrol~0.3 mmol/kg BW (Gadavist, Gadovist, BAY86-4875) — Participant received one dose of 0.3 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
  Arms: Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Drug: OptiMARK~0.1 mmol/kg BW — Participant received one dose of 0.1 mmol/kg BW of OptiMARK. OptiMARK was administered via a power injector at a rate of 2 mL/s followed by a 20 mL 0.9% saline flush at the same rate.

SUMMARY:
The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Gadavist when used for taking images of the brain and spine. The results of the MRI with Gadavist Injection will be compared to the results of MR images taken without contrast and with the results of the MR images taken with OptiMARK.

DETAILED DESCRIPTION:
Safety issues are addressed in the Adverse Events section

ELIGIBILITY:
Inclusion Criteria:

* Patients with either known or highly suspected focal areas of disruption of the blood brain barrier (BBB) (eg, primary and secondary tumors, focal inflammatory or demyelinating disorders) and/or abnormal vascularity in the CNS, who are scheduled to undergo a routine contrast-enhanced MRI of the CNS.
* Patients with untreated brain tumors should constitute a minimum of 50% of the study population and patients with treated brain tumors will be limited to a maximum of 20% of the study population

Exclusion Criteria:

* Is a female patient who is pregnant or nursing.
* Is a female of childbearing potential and did not have a negative urine pregnancy test the same day as the administration of gadobutrol or comparator treatment.
* Has received any investigational product within 30 days prior to enrolling in this study.
* Has been previously enrolled in this study or any other study using gadobutrol.
* Has any contraindication to the MRI examinations.
* Has a history of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents.
* Has received any contrast agent within 24 hours prior to gadobutrol contrast administration, or is scheduled to receive any contrast agent within 72 hours after the gadobutrol study.
* Is considered to be clinically unstable or his/her clinical course during the study period is unpredictable (eg, due to previous surgery, acute renal failure).
* Has been treated with high dose (>55 cobalt Gy equivalent) photon radiation or global radiotherapy for CNS lesions at any time before entering the study.
* Is scheduled to receive chemotherapy or radiotherapy during the study period.
* Is expected or scheduled to have a change in any treatment or procedure between the comparator and gadobutrol MRIs that may alter their interpretation.
* Is scheduled or is likely to require a biopsy or surgery within the 72 hours after the gadobutrol MRI procedure, or is scheduled for or has undergone such interventions between the comparator and gadobutrol studies.
* Has severe cardiovascular disease.
* Has any contraindication to OptiMARK according to the package insert.
* Has more than 30 brain lesions detected by any prior imaging examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- United States (20):
  - University of California Davis Medical Center, Sacramento, California
  - University of California-San Diego Medical Center, San Diego, California
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana Neuroscience Institute, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Methodist Hospital, Omaha, Nebraska
  - NYU Langone Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Argentina (2):
  - TCba Salguero, Buenos Aires, Buenos Aires
  - Fundacion Cientifica del Sur, Lornas de Zamora, Buenos Aires
- Hospital da Beneficiência Portuguesa, São Paulo, São Paulo, Brazil
- Colombia (4):
  - Centro de Diagnostico Medico, Medellín, Antioquia
  - Fundación Instituto de Alta tecnología médica de Antioquia, Medellín, Antioquia
  - DIME Clinica Neurocardiovascular S.A., Cali, Valle del Cauca Department
  - Fundación Clínica Valle del Lili, Cali

REFERENCES:
- [Derived] Breuer J, Gutierrez J, Latchaw R, Lehr R, Sorensen AG. Gadobutrol in the central nervous system at three doses: results from a phase II, randomized, multicenter trial. J Magn Reson Imaging. 2014 Feb;39(2):410-8. doi: 10.1002/jmri.24180. Epub 2013 May 16. PMID 23681501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of the first participant's first visit was 27 August 2005. The date of the last participant's last visit was 26 March 2007.
Pre-assignment Details: 242 participants were screened: 5 were screening failures (withdrew consent, did not meet study criteria, other). The remaining 237 were randomized to the 0.3, 0.1, or 0.03 millimole per kilogram (mmol/kg) group.
Groups:
- Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875): Participant received one dose of 0.03 mmol/kg body weight (BW) of Gadobutrol and one dose of 0.1 mmol/kg BW of OptiMARK. The order in which the participants received Gadobutrol and OptiMARK was randomized. Gadobutrol was administered via a power injector at a rate of 5 milliliter per second (mL/s) followed by a 20 mL 0.9% saline flush at the same rate.
Period: Overall Study
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Started | 72 | 93 | 72
Participants Received Treatment | 70 (Number reflects all treated participants of whom 67 received Gadobutrol and 70 received OptiMARK) | 90 (Number reflects all treated participants of whom 90 received Gadobutrol and 88 received OptiMARK) | 69 (Number reflects all treated participants of whom 68 received Gadobutrol and 69 received OptiMARK)
Completed | 66 | 85 | 66
Not Completed | 6 | 8 | 6
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Personal reasons | 1 | 0 | 0
Not completed — Operation | 1 | 1 | 0
Not completed — Intravenous (IV) site problems | 1 | 0 | 1
Not completed — Unable to hold still for imaging | 0 | 1 | 0
Not completed — Inclusion/exclusion criteria not met | 0 | 1 | 0
Not completed — Administrative problems | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875): Participant received one dose of 0.03 millimole per kilogram of body weight (mmol/kg BW) of Gadobutrol and one dose of 0.1 mmol/kg BW of OptiMARK. The order in which the participants received Gadobutrol and OptiMARK was randomized. Gadobutrol was administered via a power injector at a rate of 5 milliliter per second (mL/s) followed by a 20 mL 0.9% saline flush at the same rate.
- Total: Total of all reporting groups
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875) | Total
Number analyzed (Participants) | 70 | 90 | 69 | 229
Age, Customized [Number; unit: Years]
  <45 years | 36 | 42 | 29 | 107
  45-64 years | 24 | 39 | 28 | 91
  >=65 years | 10 | 9 | 12 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 58 | 38 | 129
  Male | 37 | 32 | 31 | 100
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 30 | 45 | 29 | 104
  Black | 7 | 8 | 3 | 18
  Hispanic | 3 | 6 | 3 | 12
  Asian | 1 | 1 | 0 | 2
  Other | 29 | 30 | 34 | 93

OUTCOME MEASURES:

1. Primary Outcome: Categorical Visualization Score (CVS)
Description: The primary visualization variables (number [no.] of lesions detected, border delineation, contrast enhancement, internal morphology) were condensed to a composite score (CVS). Each variable was considered a category; the CVS was calculated as: CVS=(No. of categories with increase over precontrast)-(No. of categories with decrease over precontrast). The possible outcomes of the CVS for a participant and each reader were in the range of - 3 to +4. The CVS was averaged across the 3 blinded readers, producing 1 mean CVS per participant. The higher the CVS, the more effective the treatment.
Time Frame: up to 2 hours after the injection of study medication
Population: The per protocol set (PPS), which included all participants with valid images who received +/-10% of the intended dose of study drug and had no major protocol or Magnetic Resonance Imaging (MRI) procedure deviations (excluding one participant with insufficient images)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875): Participant received one dose of 0.03 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
- Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875): Participant received one dose of 0.1 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
- Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875): Participant received one dose of 0.3 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 55 | 56
Scores on a scale | 1.43 (1.07) | 2.02 (1.04) | 1.98 (1.20)
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); 2 sample t-test between the dose groups; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = 0.59, Standard Deviation 1.49
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.844, t-test, 2 sided; Mean Difference (Final Values) = -0.04, Standard Deviation 1.59

2. Primary Outcome: Difference in Number of Lesions Detected in Pre-contrast and Combined Pre-/Post-contrast MRI.
Description: Three blinded readers evaluated the unenhanced MRI sets and the combined unenhanced/gadobutrol-enhanced MRI sets to evaluate the number of lesions, which was then averaged to produce an average reader value.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding one participant with insufficient images)
Measure: Mean (Standard Deviation); unit: Lesions per participant
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 55 | 56
Lesions per participant | -0.03 (1.82) | 0.04 (2.28) | 0.09 (2.22)
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.069, 95% CI [-0.825 to 0.69], Standard Deviation 2.92
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.53, 95% CI [-0.90 to 0.79], Standard Deviation 3.18

3. Primary Outcome: Assessment of Lesion Contrast Enhancement
Description: The blinded readers assessed the degree of contrast enhancement for each lesion on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement, which was then averaged to produce an average reader score.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no lesion detected)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 58 | 55 | 53
scores on a scale | 0.98 (0.93) | 1.78 (1.07) | 1.79 (1.15)
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.80, 95% CI [-1.17 to -0.42], Standard Deviation 1.42
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.01, 95% CI [-0.44 to 0.41], Standard Deviation 1.57

4. Primary Outcome: Assessment of Border Delineation
Description: The blinded readers assessed the delineation for each lesion on a 4-point scale where 1 = none and 4 = excellent, which was then averaged to produce an average reader score.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no lesion detected)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 58 | 55 | 53
scores on a scale | 0.28 (0.60) | 0.68 (0.61) | 0.70 (0.60)
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.40, 95% CI [-0.619 to -0.17], Standard Deviation 0.86
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.02, 95% CI [-0.25 to 0.22], Standard Deviation 1.01

5. Primary Outcome: Assessment of Internal Morphology
Description: The blinded readers assessed the degree of information available about internal morphology and structure for each lesion on a 3-point scale where 1 = poor and 3 = good, which was then averaged to produce an average reader score.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no lesion detected)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 58 | 55 | 53
scores on a scale | 0.52 (0.50) | 0.90 (0.57) | 0.80 (0.51)
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -0.38, 95% CI [-0.58 to -0.18], Standard Deviation 0.76
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = 0.10, 95% CI [-0.10 to 0.31], Standard Deviation 0.76

6. Primary Outcome: Contrast to Noise Ratio (CNR) Between White and Gray Matter With Gadobutrol Perfusion MRI
Description: CNR between white and gray matter in the perfusion imaging was defined as the signal intensity (SI) difference between white and gray matter divided by the standard deviation of the SI of white matter. An independent radiologist evaluated the gadobutrol-enhanced perfusion MRI for signal intensity.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding participants with insufficient images)
Measure: Mean (Standard Deviation); unit: CNR
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 60 | 56 | 55
CNR | 9.42 (11.4) | 27.0 (75.6) | 22.2 (15.2)
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); difference in CNR between doses and confidence interval; Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = -17.54, 95% CI [-37.11 to 2.02], Standard Deviation 76.45
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; confidence interval using t-distribution; Mean Difference (Final Values) = 4.74, 95% CI [-15.86 to 25.35], Standard Deviation 77.11

7. Secondary Outcome: Accuracy Comparison of Gadobutrol Doses - Detection of Matched Lesions: Blinded Reader 1
Description: The percent accuracy (total number of lesions matching the comparator divided by the total number of lesions identified by gadobutrol) comparison of the 0.03 and 0.1 mmol/kg gadobutrol doses and the 0.1 and 0.3 mmol/kg gadobutrol doses using detection of all comparator-detected matched lesions was performed for blinded reader (BR) 1.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no lesion detected)
Measure: Number; unit: percentage of lesions
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 60 | 56 | 55
percentage of lesions | 63.58 | 65.24 | 54.49
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.80, Chi-squared; Adjusted for clustering; accuracy difference = 1.66, 95% CI [-10.93 to 14.24], Standard Error of Mean 6.29
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.13, Chi-squared; adjusted for clustering; difference in accuracies = -10.75, 95% CI [-24.41 to 2.90], Standard Error of Mean 6.83

8. Secondary Outcome: Accuracy Comparison of Gadobutrol Doses - Detection of Matched Lesions: Blinded Reader 2
Description: The percent accuracy (total number of lesions matching the comparator divided by the total number of lesions identified by gadobutrol) comparison of the 0.03 and 0.1 mmol/kg gadobutrol doses and the 0.1 and 0.3 mmol/kg gadobutrol doses using detection of all comparator-detected matched lesions was performed for BR 2
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no lesion detected)
Measure: Number; unit: percentage of lesions
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 59 | 56 | 54
percentage of lesions | 57.62 | 71.05 | 57.47
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.03, Chi-squared; adjusted for clustering; difference in accuracy = 13.43, 95% CI [1.53 to 25.33]
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.02, Chi-squared; adjusted for clustering; difference in accuracies = -13.58, 95% CI [-25.07 to -2.09]

9. Secondary Outcome: Accuracy Comparison of Gadobutrol Doses - Detection of Matched Lesions: Blinded Reader 3
Description: The percent accuracy (total number of lesions matching the comparator divided by the total number of lesions identified by gadobutrol) comparison of the 0.03 and 0.1 mmol/kg gadobutrol doses and the 0.1 and 0.3 mmol/kg gadobutrol doses using detection of all comparator-detected matched lesions was performed for BR 3
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no lesion detected)
Measure: Number; unit: percentage of lesions
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 59 | 56 | 56
percentage of lesions | 63.31 | 57.18 | 50.05
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.11, Chi-squared; adjusted for clustering; difference in accuracy = -6.13, 95% CI [-13.73 to 1.48]
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.55, Chi-squared; adjusted for clustering; difference in accuracies = 2.87, 95% CI [-6.59 to 12.32]

10. Secondary Outcome: Accuracy Comparison of Gadobutrol Doses - Detection of Matched Enhanced Lesions: Blinded Reader 1
Description: The percent accuracy (total number of lesions matching the comparator divided by the total number of lesions identified by gadobutrol) comparison of the 0.03 and 0.1 mmol/kg gadobutrol doses and the 0.1 and 0.3 mmol/kg gadobutrol doses using detection of all comparator-detected matched enhanced lesions was performed for BR 1
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no enhanced lesion detected)
Measure: Number; unit: percentage of lesions
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 52 | 48 | 50
percentage of lesions | 48.10 | 72.73 | 55.21
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.02, Chi-squared; adjusted for clustering; difference in accuracy = 24.63, 95% CI [5.39 to 43.86]
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.13, Chi-squared; adjusted for clustering; difference in accuracy = -10.75, 95% CI [-24.41 to 2.90]

11. Secondary Outcome: Accuracy Comparison of Gadobutrol Doses - Detection of Matched Enhanced Lesions: Blinded Reader 2
Description: The percent accuracy (total number of lesions matching the comparator divided by the total number of lesions identified by gadobutrol) comparison of the 0.03 and 0.1 mmol/kg gadobutrol doses and the 0.1 and 0.3 mmol/kg gadobutrol doses using detection of all comparator-detected matched enhanced lesions was performed for BR 2
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects with no enhanced lesion detected)
Measure: Number; unit: percentage of lesions
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 47 | 44 | 44
percentage of lesions | 69.23 | 82.14 | 63.77
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.07, Chi-squared; adjusted for clustering; difference in accuracy = 12.91, 95% CI [-1.44 to 27.26]
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.02, Chi-squared; adjusted for clustering; difference in accuracy = -18.37, 95% CI [-33.60 to -1.35]

12. Secondary Outcome: Accuracy Comparison of Gadobutrol Doses - Detection of Matched Enhanced Lesions: Blinded Reader 3
Description: The percent accuracy (total number of lesions matching the comparator divided by the total number of lesions identified by gadobutrol) comparison of the 0.03 and 0.1 mmol/kg gadobutrol doses and the 0.1 and 0.3 mmol/kg gadobutrol doses using detection of all comparator-detected matched enhanced lesions was performed for BR 3
Time Frame: up to 2 hours after the injection of study medication
Population: PPS(excluding subjects with no enhanced lesion detected)
Measure: Number; unit: percentage of lesions
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 51 | 46 | 48
percentage of lesions | 55.07 | 73.53 | 68.24
Statistical Analysis 1: Comparison: Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.02, Chi-squared; adjusted for clustering; difference in accuracy = 18.46, 95% CI [3.15 to 33.77]
Statistical Analysis 2: Comparison: Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) vs Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.45, Chi-squared; adjusted for clustering; difference in accuracy = -5.29, 95% CI [-18.83 to 8.24]

13. Secondary Outcome: Evaluation of the Correct Diagnosis Following Gadobutrol-enhanced and Unenhanced MRI
Description: The gadobutrol-enhanced and unenhanced MRI diagnoses of the average reader were compared to the final diagnosis.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of exact matches
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of exact matches
  yes | 62.3 | 57.1 | 54.2
  no | 37.7 | 42.9 | 45.8

14. Secondary Outcome: Evaluation of the Diagnostic Confidence Based on Unenhanced MRI and Combined Unenhanced and Enhanced MRI
Description: The diagnostic confidence, the level of certainty in a diagnosis, was determined based on the average of the blinded readers.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS, Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  not confident | 3.3 | 3.6 | 3.6
  somewhat confident | 23.0 | 28.6 | 23.2
  confident | 49.2 | 33.9 | 39.3
  very confident | 24.6 | 33.9 | 33.9

15. Secondary Outcome: Evaluation of Perfusion Map Quality (Uncorrected Cerebral Blood Volume [CBV]) - Blinded Reader 1
Description: BR 1 evaluated the visibility of the lesion(s) on the uncorrected CBV perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS, Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Applicable (Appl.) | 8.2 | 7.1 | 3.6
  missing | 1.6 | 0 | 0
  not visible | 16.4 | 10.7 | 21.4
  poor | 21.3 | 17.9 | 12.5
  moderate | 16.4 | 19.6 | 12.5
  good | 23 | 19.6 | 17.9
  excellent | 13.1 | 25 | 32.1

16. Secondary Outcome: Evaluation of Perfusion Map Quality (Uncorrected Cerebral Blood Volume (CBV)) - Blinded Reader 2
Description: BR 2 evaluated the visibility of the lesion(s) on the uncorrected CBV perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 9.8 | 10.7 | 10.7
  missing | 1.6 | 0 | 0
  not visible | 8.2 | 12.5 | 8.9
  poor | 27.9 | 12.5 | 12.5
  moderate | 24.6 | 21.4 | 16.1
  good | 19.7 | 23.2 | 26.8
  excellent | 8.2 | 19.6 | 25

17. Secondary Outcome: Evaluation of Perfusion Map Quality (Uncorrected Cerebral Blood Volume (CBV)) - Blinded Reader 3
Description: BR 3 evaluated the visibility of the lesion(s) on the uncorrected CBV perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 11.5 | 8.9 | 16.1
  missing | 1.6 | 0 | 0
  not visible | 13.1 | 23.2 | 19.6
  poor | 23 | 12.5 | 12.5
  moderate | 26.2 | 23.2 | 16.1
  good | 16.4 | 12.5 | 10.7
  excellent | 8.2 | 19.6 | 25

18. Secondary Outcome: Evaluation of Perfusion Map Quality (Corrected Cerebral Blood Volume (CBV)) - Blinded Reader 1
Description: BR 1 evaluated the visibility of the lesion(s) on the corrected CBV perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 8.2 | 10.7 | 3.6
  missing | 1.6 | 0 | 0
  not visible | 6.6 | 14.3 | 25
  poor | 24.6 | 19.6 | 10.7
  moderate | 21.3 | 8.9 | 8.9
  good | 19.7 | 21.4 | 30.4
  excellent | 18 | 25 | 21.4

19. Secondary Outcome: Evaluation of Perfusion Map Quality (Corrected Cerebral Blood Volume (CBV)) - Blinded Reader 2
Description: BR 2 evaluated the visibility of the lesion(s) on the corrected CBV perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 11.5 | 16.1 | 7.1
  missing | 1.6 | 0 | 0
  not visible | 6.6 | 5.4 | 14.3
  poor | 21.3 | 14.3 | 7.1
  moderate | 23 | 21.4 | 14.3
  good | 26.2 | 17.9 | 32.1
  excellent | 9.8 | 25 | 25

20. Secondary Outcome: Evaluation of Perfusion Map Quality (Corrected Cerebral Blood Volume (CBV)) - Blinded Reader 3
Description: BR 3 evaluated the visibility of the lesion(s) on the corrected CBV perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 11.5 | 12.5 | 17.9
  missing | 1.6 | 1.8 | 0
  not visible | 14.8 | 19.6 | 23.2
  poor | 24.6 | 12.5 | 10.7
  moderate | 19.7 | 17.9 | 10.7
  good | 21.3 | 16.1 | 23.2
  excellent | 6.6 | 19.6 | 14.3

21. Secondary Outcome: Evaluation of Perfusion Map Quality (Cerebral Blood Flow (CBF)) - Blinded Reader 1
Description: BR 1 evaluated the visibility of the lesion(s) on the CBF perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 6.6 | 12.5 | 1.8
  missing | 1.6 | 0 | 0
  not visible | 13.1 | 14.3 | 23.2
  poor | 31.1 | 7.1 | 14.3
  moderate | 14.8 | 17.9 | 12.5
  good | 9.8 | 17.9 | 30.4
  excellent | 23 | 30.4 | 17.9

22. Secondary Outcome: Evaluation of Perfusion Map Quality (Cerebral Blood Flow (CBF)) - Blinded Reader 2
Description: BR 2 evaluated the visibility of the lesion(s) on the CBF perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 8.2 | 12.5 | 8.9
  missing | 1.6 | 0 | 0
  not visible | 11.5 | 12.5 | 12.5
  poor | 21.3 | 8.9 | 19.6
  moderate | 23 | 25 | 25
  good | 24.6 | 16.1 | 8.9
  excellent | 9.8 | 25 | 25

23. Secondary Outcome: Evaluation of Perfusion Map Quality (Cerebral Blood Flow (CBF)) - Blinded Reader 3
Description: BR 3 evaluated the visibility of the lesion(s) on the CBF perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 13.1 | 10.7 | 16.1
  missing | 1.6 | 1.8 | 0
  not visible | 14.8 | 17.9 | 25
  poor | 14.8 | 21.4 | 12.5
  moderate | 31.1 | 10.7 | 10.7
  good | 18 | 19.6 | 17.9
  excellent | 6.6 | 17.9 | 17.9

24. Secondary Outcome: Evaluation of Perfusion Map Quality (Time to Peak (TTP)) - Blinded Reader 1
Description: BR 1 evaluated the visibility of the lesion(s) on the TTP perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 6.6 | 8.9 | 5.4
  missing | 1.6 | 1.8 | 0
  not visible | 34.4 | 21.4 | 26.8
  poor | 29.5 | 14.3 | 21.4
  moderate | 9.8 | 10.7 | 10.7
  good | 13.1 | 17.9 | 14.3
  excellent | 4.9 | 25 | 21.4

25. Secondary Outcome: Evaluation of Perfusion Map Quality (Time to Peak (TTP)) - Blinded Reader 2
Description: BR 2 evaluated the visibility of the lesion(s) on the TTP perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 24.6 | 17.9 | 8.9
  missing | 1.6 | 0 | 0
  not visible | 18 | 5.4 | 14.3
  poor | 26.2 | 21.4 | 30.4
  moderate | 11.5 | 33.9 | 23.2
  good | 13.1 | 17.9 | 17.9
  excellent | 4.9 | 3.6 | 5.4

26. Secondary Outcome: Evaluation of Perfusion Map Quality (Time to Peak (TTP)) - Blinded Reader 3
Description: BR 3 evaluated the visibility of the lesion(s) on the TTP perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 11.5 | 10.7 | 17.9
  missing | 1.6 | 1.8 | 0
  not visible | 32.8 | 25 | 21.4
  poor | 23 | 23.2 | 16.1
  moderate | 18 | 19.6 | 25
  good | 9.8 | 16.1 | 10.7
  excellent | 3.3 | 3.6 | 8.9

27. Secondary Outcome: Evaluation of Perfusion Map Quality (Mean Transit Time (MTT)) - Blinded Reader 1
Description: BR 1 evaluated the visibility of the lesion(s) on the MTT perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 8.2 | 7.1 | 3.6
  missing | 1.6 | 0 | 0
  not visible | 16.4 | 16.1 | 19.6
  poor | 19.7 | 19.6 | 19.6
  moderate | 26.2 | 12.5 | 14.3
  good | 19.7 | 26.8 | 25
  excellent | 8.2 | 17.9 | 17.9

28. Secondary Outcome: Evaluation of Perfusion Map Quality (Mean Transit Time (MTT)) - Blinded Reader 2
Description: BR 2 evaluated the visibility of the lesion(s) on the MTT perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 13.1 | 16.1 | 12.5
  missing | 1.6 | 0 | 0
  not visible | 14.8 | 14.3 | 14.3
  poor | 37.7 | 30.4 | 23.2
  moderate | 16.4 | 16.1 | 17.9
  good | 13.1 | 12.5 | 19.6
  excellent | 3.3 | 10.7 | 12.5

29. Secondary Outcome: Evaluation of Perfusion Map Quality (Mean Transit Time (MTT)) - Blinded Reader 3
Description: BR 3 evaluated the visibility of the lesion(s) on the MTT perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 11.5 | 12.5 | 16.1
  missing | 1.6 | 1.8 | 0
  not visible | 19.7 | 25 | 21.4
  poor | 19.7 | 12.5 | 16.1
  moderate | 29.5 | 30.4 | 12.5
  good | 13.1 | 7.1 | 17.9
  excellent | 4.9 | 10.7 | 16.1

30. Secondary Outcome: Evaluation of Perfusion Map Quality (Permeability Factor (PF) - Blinded Reader 1
Description: BR 1 evaluated the visibility of the lesion(s) on the PF perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 13.1 | 8.9 | 1.8
  not visible | 11.5 | 21.4 | 28.6
  poor | 21.3 | 23.2 | 19.6
  moderate | 13.1 | 7.1 | 17.9
  good | 19.7 | 21.4 | 17.9
  excellent | 21.3 | 17.9 | 14.3

31. Secondary Outcome: Evaluation of Perfusion Map Quality (Permeability Factor (PF) - Blinded Reader 2
Description: BR 2 evaluated the visibility of the lesion(s) on the PF perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS. Due to rounding, the sum of the percentages may range from 99.9 to 100.1.
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 14.8 | 16.1 | 8.9
  missing | 3.3 | 0 | 0
  not visible | 6.6 | 14.3 | 16.1
  poor | 21.3 | 17.9 | 16.1
  moderate | 26.2 | 28.6 | 25
  good | 19.7 | 16.1 | 26.8
  excellent | 8.2 | 7.1 | 7.1

32. Secondary Outcome: Evaluation of Perfusion Map Quality (Permeability Factor (PF)) - Blinded Reader 3
Description: BR 3 evaluated the visibility of the lesion(s) on the PF perfusion map.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Not Appl. | 11.5 | 10.7 | 19.6
  missing | 4.9 | 3.6 | 0
  not visible | 13.1 | 26.8 | 25
  poor | 24.6 | 14.3 | 14.3
  moderate | 21.3 | 12.5 | 12.5
  good | 18 | 21.4 | 17.9
  excellent | 6.6 | 10.7 | 10.7

33. Secondary Outcome: Evaluation of Perfusion Map Parameter Value (Uncorrected Cerebral Blood Volume (CBV)) - Independent Radiologist
Description: The independent radiologist determined the uncorrected CBV for each lesion. CBV is the volume of blood in the tissue.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects whose parameter map value was not determined)
Measure: Mean (Standard Deviation); unit: mL / 100 g tissue
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 55 | 45 | 42
mL / 100 g tissue | 114.61 (127.75) | 346.81 (313.49) | 1209.89 (1121.63)

34. Secondary Outcome: Evaluation of Perfusion Map Parameter Value (Corrected Cerebral Blood Volume (CBV)) - Independent Radiologist
Description: The independent radiologist determined the corrected CBV for each lesion. CBV is the volume of blood in the tissue.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects whose parameter map value was not determined)
Measure: Mean (Standard Deviation); unit: mL / 100 g tissue
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 55 | 44 | 42
mL / 100 g tissue | 2728.71 (2788.59) | 2682.97 (1493.95) | 3382.20 (1908.56)

35. Secondary Outcome: Evaluation of Perfusion Map Parameter Value (Cerebral Blood Flow (CBF)) - Independent Radiologist
Description: The independent radiologist determined the CBF for each lesion. CBF is the volume of blood passing through tissue per unit of time.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects whose parameter map value was not determined)
Measure: Mean (Standard Deviation); unit: mL / 100 g tissue / min.
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 55 | 44 | 42
mL / 100 g tissue / min. | 4.80 (6.37) | 5.15 (4.30) | 3.48 (2.24)

36. Secondary Outcome: Evaluation of Perfusion Map Parameter Value (Time to Peak (TTP)) - Independent Radiologist
Description: The independent radiologist determined the TTP for each lesion. TTP is the delay between the arrival of the contrast agent bolus arrival time and the peak of the concentration curve.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects whose parameter map value was not determined)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 55 | 45 | 42
seconds | 79.39 (25.43) | 80.31 (27.21) | 86.52 (28.70)

37. Secondary Outcome: Evaluation of Perfusion Map Parameter Value (Mean Transit Time (MTT)) - Independent Radiologist
Description: The independent radiologist determined the MTT for each lesion. The MTT is the time (seconds) for contrast to pass through tissues.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects whose parameter map value was not determined)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 55 | 44 | 42
seconds | 6.30 (4.77) | 6.02 (3.71) | 7.05 (4.54)

38. Secondary Outcome: Evaluation of Perfusion Map Parameter Value (Permeability Factor (PF)) - Independent Radiologist
Description: The independent radiologist determined the PF for each lesion
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects whose parameter map value was not determined)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 54 | 44 | 42
seconds | 4.04 (3.35) | 1.65 (0.82) | 0.99 (1.88)

39. Secondary Outcome: Evaluation of Perfusion Map Artifacts (Uncorrected Cerebral Blood Volume (CBV)) - Blinded Reader
Description: The blinded reader evaluated if artifacts were present on the uncorrected CBV perfusion map and recorded the type of the major artifact. EPI: echo-planar imaging; T2: transversal relaxation time.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Blinded Reader 1 - Missing | 1.6 | 0 | 0
  Blinded Reader 1 - 0 none | 72.1 | 75 | 69.6
  Blinded Reader 1 - EPI distortion | 24.6 | 23.2 | 21.4
  Blinded Reader 1 - movement artifacts | 0 | 0 | 1.8
  Blinded Reader 1 - other | 1.6 | 1.8 | 7.1
  Blinded reader 2 - Missing | 1.6 | 0 | 0
  Blinded Reader 2 - 0 none | 62.3 | 66.1 | 89.3
  Blinded Reader 2 - EPI distortion | 3.3 | 10.7 | 5.4
  Blinded Reader 2 - movement artifacts | 32.8 | 23.2 | 3.6
  Blinded Reader 2 - other | 0 | 0 | 1.8
  Blinded Reader 3 - Missing | 1.6 | 0 | 0
  Blinded Reader 3 - none | 62.3 | 67.9 | 78.6
  Blinded Reader 3 - EPI distortion | 6.6 | 16.1 | 10.7
  Blinded Reader 3 - T2 artifacts | 3.3 | 10.7 | 3.6
  Blinded Reader 3 - movement artifacts | 14.8 | 3.6 | 3.6
  Blinded Reader 3 - other | 11.5 | 1.8 | 3.6

40. Secondary Outcome: Evaluation of Perfusion Map Artifacts (Corrected Cerebral Blood Volume (CBV)) - Blinded Reader
Description: The blinded reader evaluated if artifacts were present on the corrected CBV perfusion map and recorded the type of the major artifact. EPI: echo-planar imaging; T2: transversal relaxation time. CBV is the fraction of the tissue volume occupied by the blood.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Blinded Reader 1 - Missing | 1.6 | 0 | 0
  Blinded Reader 1 - 0 none | 75.4 | 76.8 | 66.1
  Blinded Reader 1 - EPI distortion | 21.3 | 23.2 | 28.6
  Blinded Reader 1 - other | 1.6 | 0 | 5.4
  Blinded Reader 2 - Missing | 1.6 | 0 | 0
  Blinded Reader 2 - 0 none | 78.7 | 80.4 | 83.9
  Blinded Reader 2 - EPI distortion | 6.6 | 8.9 | 14.3
  Blinded Reader 2 - movement artifacts | 13.1 | 10.7 | 0
  Blinded Reader 2 - other | 0 | 0 | 1.8
  Blinded Reader 3 - Missing | 1.6 | 1.8 | 0
  Blinded Reader 3 - 0 none | 55.7 | 69.6 | 76.8
  Blinded Reader 3 - EPI distortion | 4.9 | 12.5 | 12.5
  Blinded Reader 3 - T2 artifacts | 6.6 | 10.7 | 3.6
  Blinded Reader 3 - movement artifacts | 23 | 1.8 | 1.8
  Blinded Reader 3 - other | 8.2 | 3.6 | 5.4

41. Secondary Outcome: Evaluation of Perfusion Map Artifacts (Cerebral Blood Flow (CBF)) - Blinded Reader
Description: The blinded reader evaluated if artifacts were present on the CBF perfusion map and recorded the type of the major artifact. EPI: echo-planar imaging; T2: transversal relaxation time
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Blinded Reader 1 - Missing | 1.6 | 0 | 0
  Blinded Reader 1 - 0 none | 70.5 | 85.7 | 71.4
  Blinded Reader 1 - EPI distortion | 26.2 | 12.5 | 23.2
  Blinded Reader 1 - T2 artifacts | 1.6 | 0 | 0
  Blinded Reader 1 - other | 0 | 1.8 | 5.4
  Blinded Reader 2- Missing | 1.6 | 0 | 0
  Blinded Reader 2- 0 none | 77 | 82.1 | 80.4
  Blinded Reader 2 - EPI distortion | 6.6 | 7.1 | 10.7
  Blinded Reader 2- movement artifacts | 14.8 | 10.7 | 7.1
  Blinded Reader 2- other | 0 | 0 | 1.8
  Blinded Reader 3 - Missing | 1.6 | 1.8 | 0
  Blinded Reader 3 - 0 none | 68.9 | 76.8 | 75
  Blinded Reader 3 - EPI distortion | 6.6 | 10.7 | 12.5
  Blinded Reader 3 - T2 artifacts | 11.5 | 8.9 | 8.9
  Blinded Reader 3 - movement artifacts | 3.3 | 1.8 | 0
  Blinded Reader 3 - other | 8.2 | 0 | 3.6

42. Secondary Outcome: Evaluation of Perfusion Map Artifacts (Time to Peak (TTP)) - Blinded Reader
Description: The blinded reader evaluated if artifacts were present on the TTP perfusion map and recorded the type of the major artifact. EPI: echo-planar imaging; T2: transversal relaxation time
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Blinded Reader 1 - missing | 1.6 | 1.8 | 0
  Blinded Reader 1 - 0 none | 75.4 | 76.8 | 75
  Blinded Reader 1 - EPI distortion | 14.8 | 21.4 | 19.6
  Blinded Reader 1- movement artifacts | 1.6 | 0 | 0
  Blinded Reader 1 - other | 6.6 | 0 | 5.4
  Blinded Reader 2 - missing | 1.6 | 0 | 0
  Blinded Reader 2 - 0 none | 34.4 | 62.5 | 71.4
  Blinded Reader 2 - EPI distortion | 6.6 | 8.9 | 10.7
  Blinded Reader 2 - movement artifacts | 37.7 | 19.6 | 17.9
  Blinded Reader 2 - other | 19.7 | 8.9 | 0
  Blinded Reader 3 - missing | 1.6 | 1.8 | 0
  Blinded Reader 3 - 0 none | 41 | 57.1 | 64.3
  Blinded Reader 3 - EPI distortions | 4.9 | 10.7 | 12.5
  Blinded Reader 3 - T2 artifacts | 3.3 | 8.9 | 8.9
  Blinded Reader3 - movement artifacts | 26.2 | 5.4 | 7.1
  Blinded Reader 3 - other | 23 | 16.1 | 7.1

43. Secondary Outcome: Evaluation of Perfusion Map Artifacts (Mean Transit Time (MTT)) - Blinded Reader
Description: The blinded reader evaluated if artifacts were present on the MTT perfusion map and recorded the type of the major artifact. EPI: echo-planar imaging; T2: transversal relaxation time
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Blinded Reader 1 - missing | 1.6 | 0 | 0
  Blinded Reader 1 - 0 none | 80.3 | 67.9 | 71.4
  Blinded Reader 1 - EPI distortion | 16.4 | 30.4 | 19.6
  Blinded Reader 1 - T2 artifacts | 0 | 0 | 1.8
  Blinded Reader 1 - movement artifacts | 0 | 0 | 1.8
  Blinded Reader 1 - other | 1.6 | 1.8 | 5.4
  Blinded Reader 2 - missing | 1.6 | 0 | 0
  Blinded Reader 2 - none | 41 | 71.4 | 73.2
  Blinded Reader 2 - EPI distortion | 1.6 | 5.4 | 8.9
  Blinded Reader 2 - movement artifacts | 52.5 | 23.2 | 16.1
  Blinded Reader 2 - other | 3.3 | 0 | 1.8
  Blinded Reader 3 - missing | 1.6 | 1.8 | 0
  Blinded Reader 3 - 0 none | 50.8 | 66.1 | 69.6
  Blinded Reader 3 - EPI distortion | 8.2 | 7.1 | 16.1
  Blinded Reader 3 - T2 artifacts | 3.3 | 5.4 | 5.4
  Blinded Reader 3 - movement artifacts | 26.2 | 10.7 | 5.4
  Blinded Reader 3 - other | 9.8 | 8.9 | 3.6

44. Secondary Outcome: Evaluation of Perfusion Map Artifacts (Permeability Factor (PF)) - Blinded Reader
Description: The blinded reader evaluated if artifacts were present on the PF perfusion map and recorded the type of the major artifact. EPI: echo-planar imaging; T2: transversal relaxation time
Time Frame: up to 2 hours after the injection of study medication
Population: PPS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 56 | 56
percentage of participants
  Blinded Reader 1 - 0 none | 73.8 | 75 | 71.4
  Blinded Reader 1 - EPI distortion | 21.3 | 23.2 | 26.8
  Blinded Reader 1 - T2 artifacts | 0 | 1.8 | 0
  Blinded Reader 1 - movement artifacts | 1.6 | 0 | 0
  Blinded Reader 1 - other | 3.3 | 0 | 1.8
  Blinded Reader 2 - missing | 3.3 | 0 | 0
  Blinded Reader 2 - 0 none | 73.8 | 75 | 73.2
  Blinded Reader 2 - EPI distortion | 4.9 | 8.9 | 12.5
  Blinded Reader 2 - movement artifacts | 16.4 | 16.1 | 14.3
  Blinded Reader 2 - other | 1.6 | 0 | 0
  Blinded Reader 3 - missing | 4.9 | 3.6 | 0
  Blinded Reader 3 - 0 none | 37.7 | 51.8 | 69.6
  Blinded Reader 3 - EPI distortion | 8.2 | 10.7 | 12.5
  Blinded Reader 3 - T2 artifacts | 4.9 | 10.7 | 5.4
  Blinded Reader 3 - movement artifacts | 36.1 | 14.3 | 7.1
  Blinded Reader 3 - other | 8.2 | 8.9 | 5.4

45. Secondary Outcome: Evaluation of MRI Tumor Grade Agreement With Biopsy Results by Dose Group
Description: The blinded readers gave an estimation of the tumor grade of brain tumors (low grade [I or II] or high grade [III or IV]) in terms of malignancy using the information obtained by perfusion imaging, which was compared to the biopsy sample results
Time Frame: up to 2 hours after the injection of study medication
Population: PPS participants with tumors
Measure: Number; unit: Percentage of accuracy
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 61 | 55 | 56
Percentage of accuracy
  Blinded Reader 1 | 60.0 | 57.1 | 40.0
  Blinded Reader 2 | 40.0 | 42.9 | 40.0
  Blinded Reader 3 | 60.0 | 57.1 | 30.0

46. Secondary Outcome: Contrast to Noise Ratio (CNR) of Lesion/Gray Matter and Lesion/White Matter
Description: CNR between lesion/gray matter and lesion/white matter in the perfusion imaging was defined as the signal intensity (SI) difference between lesion and gray or white matter divided by the standard deviation of background noise. An independent radiologist evaluated the gadobutrol-enhanced perfusion MRI for signal intensity.
Time Frame: up to 2 hours after the injection of study medication
Population: PPS (excluding subjects who had no lesion detected, and those who had no value determined)
Measure: Mean (Standard Deviation); unit: CNR
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 48 | 44 | 39
CNR
  lesion gray | -0.03 (13.0) | 13.0 (78.4) | 5.38 (25.0)
  lesion white | -10 (12) | -17 (19.9) | -17 (20.4)

ADVERSE EVENTS:
Groups:
- Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875): Reporting Group 1 (RG1): Participant received one dose of 0.03 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
- Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875): Reporting group 2 (RG2): Participant received one dose of 0.1 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
- Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875): Reporting group 3 (RG3): Participant received one dose of 0.3 mmol/kg BW of Gadobutrol. Gadobutrol was administered via a power injector at a rate of 5 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
- Optimark~0.1mmol/kg BW: Reporting group 4 (RG4): Participant received one dose of 0.1 mmol/kg BW of OptiMARK. OptiMARK was administered via a power injector at a rate of 2 mL/s followed by a 20 mL 0.9% saline flush at the same rate.
Arm/Group | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875) | Optimark~0.1mmol/kg BW
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/90 | 0/68 | 1/227
Other Adverse Events (participants affected / at risk) | 19/67 | 30/90 | 22/68 | 23/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) (N=67) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) (N=90) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875) (N=68) | Optimark~0.1mmol/kg BW (N=227)
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol~0.03 mmol/kg BW (Gadavist, BAY86-4875) (N=67) | Gadobutrol~0.1 mmol/kg BW (Gadavist, BAY86-4875) (N=90) | Gadobutrol~0.3 mmol/kg BW (Gadavist, BAY86-4875) (N=68) | Optimark~0.1mmol/kg BW (N=227)
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 3
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Application site erythema (General disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 2
Injection site irritation (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 4
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 8 | 7 | 3 | 8
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 2
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0
Claustrophobia (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hyperaemia (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
OptiMARK was used as a standard of reference in this study. A formal comparison of the efficacy of gadobutrol and OptiMARK was not specified prospectively in the statistical analysis plan. For completeness, the safety data of OptiMARK is presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of results will be a group publication. Sites with recruitment of >= 6 valid patients will contribute. There will be one author from each site having contributed >= 6 valid patients. Authorship listed according to recruitment. Sponsor will appoint up to 3 persons as co-authors. Main author of publication may be announced by site with most valid patients enrolled. In case more than 1 center reaches maximum patient No., main author will be from the center with fastest recruitment